CLINICAL TRIAL: NCT06418529
Title: Comparative Effectiveness of New Initiators of Tofacitinib and Other Biologic/Targeted Synthetic DMARDs in Patients With Rheumatoid Arthritis
Brief Title: A Study to Understand How Effective is Tofacitinib When Compared to Other Advanced Treatments in Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921445; NCT06418529 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Results first posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib; Tumor Necrosis Factor Inhibitors; Abatacept; tocilizumab; sarilumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- rheumatoid arthritis: Patients diagnosed with rheumatoid arthritis
  Interventions: Drug: tofacitinib; Drug: tumor necrosis factor inhibitors (TNFi); Drug: abatacept; Drug: tocilizumab or sarilumab

INTERVENTIONS:
Drug: tofacitinib — New index treatment of tofacitinib
Drug: tumor necrosis factor inhibitors (TNFi) — New index treatment of TNFi
Drug: abatacept — New index treatment of abatacept
Drug: tocilizumab or sarilumab — New index treatment of tocilizumab or sarilumab

SUMMARY:
The purpose of this study is to learn how different types of medicines may improve disease activity in people with rheumatoid arthritis (RA). RA is a kind of joint disease that causes pain and swelling.

The study will look at data from a large, US-based group of RA patients who have taken the below medicines:

* Tofacitinib
* Abatacept
* Tocilizumab or sarilumab

The study will compare clinical disease activity scores of patients on the different medicines taken. The study will also decide whether some patient traits or disease factors play a role in how medicines may improve disease activity.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years on the cohort entry date.
2. Diagnosed with rheumatoid arthritis (RA) at any time prior to cohort entry date:

   1. At least two RA diagnosis codes at least 30 days apart, each coming from an encounter with a rheumatologist;
   2. At least one inpatient visit with a RA diagnosis code;
   3. At least two outpatient records with a RA diagnosis code at least 30 days apart and within a year, regardless of physician specialty; or
   4. At least one outpatient record with an RA diagnosis and a prescription or fill for a disease modifying anti-rheumatic drug (DMARD) from a specified list and does not have any of the non-RA conditions for which those drugs may also be prescribed.
3. Initiation of specified biologic or targeted synthetic molecule DMARDs of interest for treatment of RA (ie, tofacitinib, etanercept, adalimumab, certolizumab, golimumab, infliximab, abatacept, tocilizumab, or sarilumab).
4. At least 180 days of baseline data available prior to and including the cohort entry date.
5. At least one Clinical Disease Activity Index (CDAI) score in 45 days prior to and including the cohort entry date (baseline).

Exclusion Criteria:

1. Patients diagnosed with concomitant indications for tofacitinib [psoriatic arthritis (PsA), UC, and polyarticular course juvenile idiopathic arthritis (pcJIA)] at any time prior to cohort entry date, determined by at least two (2) diagnosis codes at least 30 days apart and prior to baseline.
2. Patients with >1 b/tsDMARD (ie, tofacitinib, etanercept, adalimumab, certolizumab, golimumab, infliximab, abatacept tocilizumab, or sarilumab) prescribed on index date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A retrospective design will be used to explore the comparative effectiveness of tofacitinib among a cohort of patients with rheumatoid arthritis (RA) in the U.S. using the OM1 PremiOM™ RA dataset (OM1, Inc., Boston, MA). This dataset of over 244,000 patients with RA is derived from deterministically linked, de-identified, individual-level healthcare claims and electronic medical record (EMR) data. EMR data are derived from several healthcare systems and rheumatologist's EMR provider systems geographically representative of the U.S. population. For this analysis, the OM1 PremiOM™ RA dataset will include the time period from 01 January 2013 through 31 December 2023.
Sampling Method: Probability Sample
Enrollment: 21340 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921445

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible retrospective data retrieved from US based OM1 PremiOM™ Rheumatoid Arthritis (RA)dataset (OM1, Inc., Boston, MA) from 1 Jan 2013 to 13 Mar 2024 (approximately 11.2 years). Dataset included participants diagnosed with RA in routine clinical care among network of rheumatologists across US. Participants who initiated treatment with tofacitinib or comparator (tumor necrosis factor inhibitor [TNFi], abatacept, interleukin 6 [IL-6]) were assigned to respective reporting groups for analysis.
Pre-assignment Details: Retrospective data retrieved, were assembled in this study from 15-May-2024 to 19-July-2024 (approximately 2 months).
Groups:
- Tofacitinib: Participants diagnosed with RA and who initiated treatment with tofacitinib, in routine clinical care in a network of rheumatologists across the US were included. Their data was observed from the date after treatment initiation until the occurrence of an outcome or a censoring event: (i) discontinued their index treatment, (ii) switched to a different targeted synthetic/biologic (ts/b)DMARD, (iii) were lost to follow-up, or (iv) on the last day of the outcome assessment window for each analysis, whichever occurred first, from 1 January 2013 to 13 March 2024 (approximately 11.2 years). Retrospective data retrieved, were assembled in this study from 15-May-2024 to 19-July-2024 (approximately 2 months). There was no study intervention administration under this study.
- TNFi: Participants diagnosed with RA and who initiated treatment with TNFi, in routine clinical care in a network of rheumatologists across the US were included. Their data was observed from the date after treatment initiation until the occurrence of an outcome or a censoring event: (i) discontinued their index treatment, (ii) switched to a different ts/bDMARD, (iii) were lost to follow-up, or (iv) on the last day of the outcome assessment window for each analysis, whichever occurred first, from 1 January 2013 to 13 March 2024 (approximately 11.2 years). Retrospective data retrieved, were assembled in this study from 15-May-2024 to 19-July-2024 (approximately 2 months). There was no study intervention administration under this study.
- Abatacept: Participants diagnosed with RA and who initiated treatment with abatacept, in routine clinical care in a network of rheumatologists across the US were included. Their data was observed from the date after treatment initiation until the occurrence of an outcome or a censoring event: (i) discontinued their index treatment, (ii) switched to a different ts/bDMARD, (iii) were lost to follow-up, or (iv) on the last day of the outcome assessment window for each analysis, whichever occurred first, from 1 January 2013 to 13 March 2024 (approximately 11.2 years). Retrospective data retrieved, were assembled in this study from 15-May-2024 to 19-July-2024 (approximately 2 months). There was no study intervention administration under this study.
- IL-6: Participants diagnosed with RA and who initiated treatment with IL-6, in routine clinical care in a network of rheumatologists across the US were included. Their data was observed from the date after treatment initiation until the occurrence of an outcome or a censoring event: (i) discontinued their index treatment, (ii) switched to a different ts/bDMARD, (iii) were lost to follow-up, or (iv) on the last day of the outcome assessment window for each analysis, whichever occurred first, from 1 January 2013 to 13 March 2024 (approximately 11.2 years). Retrospective data retrieved, were assembled in this study from 15-May-2024 to 19-July-2024 (approximately 2 months). There was no study intervention administration under this study.
Period: Overall Study
Arm/Group | Tofacitinib | TNFi | Abatacept | IL-6
Started | 3681 | 11667 | 3528 | 2464
Completed | 3681 | 11667 | 3528 | 2464
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data were retrieved from dataset and observed retrospectively in this study.
Groups:
- Tofacitinib: Participants diagnosed with RA and who initiated treatment with tofacitinib, in routine clinical care in a network of rheumatologists across the US were included. Their data was observed from the date after treatment initiation until the occurrence of an outcome or a censoring event: (i) discontinued their index treatment, (ii) switched to a different ts/bDMARD, (iii) were lost to follow-up, or (iv) on the last day of the outcome assessment window for each analysis, whichever occurred first, from 1 January 2013 to 13 March 2024 (approximately 11.2 years). Retrospective data retrieved, were assembled in this study from 15-May-2024 to 19-July-2024 (approximately 2 months). There was no study intervention administration under this study.
- Total: Total of all reporting groups
Arm/Group | Tofacitinib | TNFi | Abatacept | IL-6 | Total
Number analyzed (Participants) | 3681 | 11667 | 3528 | 2464 | 21340
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.9 (12.3) | 58.1 (13.7) | 61.1 (13.1) | 60.5 (12.8) | 59.4 (13.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2997 | 9171 | 2,898 | 1,982 | 17048
  Male | 684 | 2496 | 630 | 482 | 4292
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 210 | 639 | 172 | 134 | 1155
  Not Hispanic or Latino | 3182 | 10026 | 3,091 | 2151 | 18450
  Unknown or Not Reported | 289 | 1002 | 265 | 179 | 1735
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 330 | 1131 | 349 | 238 | 2048
  Race: White | 2776 | 8436 | 2659 | 1855 | 15726
  Race: Other | 412 | 1362 | 351 | 272 | 2397
  Race: Unknown | 163 | 738 | 169 | 99 | 1169

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Low Disease Activity (LDA) or Remission Based on Clinical Disease Activity Index (CDAI) at 6-Months Follow-up: Tofacitinib vs. TNFi
Description: CDAI is a simplified index for assessing disease activity. CDAI is the numerical sum of 4 outcome parameters: swollen joint counts (SJC) and tender/painful joint counts (TJC) (score range from 0 to 28, higher scores = worse condition), participant's global assessment of disease activity (PtGA) and physician's global assessment of disease activity (PGA) (assessed on 0-10 centimeter [cm)] visual analog scale [VAS]; higher scores = greater affection due to disease activity). CDAI total score = 0 (no disease) to 76 (severe disease), higher scores indicated worse condition. LDA was defined as CDAI score of 2.9 to 10.0 and remission was defined as CDAI score of 0.0 to 2.8. Incidence rate was defined as the number of events (LDA or remission based on CDAI score) divided by the Participant-Year, multiplied by 1000. Inverse probability of treatment weighting (IPTW) using stabilized weights to adjust for baseline confounders, was used for analysis.
Time Frame: During 6 month of follow-up post-initiation of tofacitinib or TNFi; retrospective data retrieved, were assembled in this study from 15-May-2024 to 19-July-2024 (approximately 2 months)
Population: Analysis population included all eligible participants whose data were retrieved from dataset and observed in this retrospective observational study.
Measure: Number; unit: Events per 1000 person years
Arm/Group | Tofacitinib | TNFi
Number analyzed (Participants) | 3681 | 11667
Events per 1000 person years | 426.8 | 471.9
Statistical Analysis 1: Comparison: Tofacitinib vs TNFi; Test type: Other; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.85 to 1.05]

2. Primary Outcome: Incidence Rate of LDA or Remission Based on CDAI at 12-Months Follow-up: Tofacitinib vs. TNFi
Description: CDAI is a simplified index for assessing disease activity. CDAI is the numerical sum of 4 outcome parameters: SJC and TJC (score range from 0 to 28, higher scores = worse condition), PtGA and PGA (assessed on 0-10 cm) VAS; higher scores = greater affection due to disease activity). CDAI total score = 0 (no disease) to 76 (severe disease), higher scores indicated worse condition. LDA was defined as CDAI score of 2.9 to 10.0 and remission was defined as CDAI score of 0.0 to 2.8. Incidence rate was defined as the number of events (LDA or remission based on CDAI score) divided by the Participant-Year, multiplied by 1000. IPTW using stabilized weights to adjust for baseline confounders, was used for analysis.
Time Frame: During 12 month of follow-up post-initiation of tofacitinib or TNFi; retrospective data retrieved, were assembled in this study from 15-May-2024 to 19-July-2024 (approximately 2 months)
Population: as for outcome 1
Measure: Number; unit: Events per 1000 person years
Arm/Group | Tofacitinib | TNFi
Number analyzed (Participants) | 3681 | 11667
Events per 1000 person years | 185.5 | 200.4
Statistical Analysis 1: Comparison: Tofacitinib vs TNFi; Test type: Other; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.83 to 1.07]

3. Primary Outcome: Incidence Rate of LDA or Remission Based on CDAI at 6-Months Follow-up: Tofacitinib vs. Abatacept
Description: as for outcome 2
Time Frame: During 6 month of follow-up post-initiation of tofacitinib or abatacept; retrospective data retrieved, were assembled in this study from 15-May-2024 to 19-July-2024 (approximately 2 months)
Population: as for outcome 1
Measure: Number; unit: Events per 1000 person years
Arm/Group | Tofacitinib | Abatacept
Number analyzed (Participants) | 3681 | 3528
Events per 1000 person years | 421.1 | 486.6
Statistical Analysis 1: Comparison: Tofacitinib vs Abatacept; Test type: Other; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.79 to 0.99]

4. Primary Outcome: Incidence Rate of LDA or Remission Based on CDAI at 12-Months Follow-up: Tofacitinib vs. Abatacept
Description: as for outcome 2
Time Frame: During 12 month of follow-up post-initiation of tofacitinib or abatacept; retrospective data retrieved, were assembled in this study from 15-May-2024 to 19-July-2024 (approximately 2 months)
Population: as for outcome 1
Measure: Number; unit: Events per 1000 person years
Arm/Group | Tofacitinib | Abatacept
Number analyzed (Participants) | 3681 | 3528
Events per 1000 person years | 185.2 | 203.1
Statistical Analysis 1: Comparison: Tofacitinib vs Abatacept; Test type: Other; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.79 to 1.04]

5. Primary Outcome: Incidence Rate of LDA or Remission Based on CDAI at 6-Months Follow-up: Tofacitinib vs. IL-6
Description: as for outcome 2
Time Frame: During 6 month of follow-up post-initiation of tofacitinib or IL-6; retrospective data retrieved, were assembled in this study from 15-May-2024 to 19-July-2024 (approximately 2 months)
Population: as for outcome 1
Measure: Number; unit: Events per 1000 person years
Arm/Group | Tofacitinib | IL-6
Number analyzed (Participants) | 3681 | 2464
Events per 1000 person years | 401.7 | 436.3
Statistical Analysis 1: Comparison: Tofacitinib vs IL-6; Test type: Other; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.81 to 1.05]

6. Primary Outcome: Incident Rate of Low Disease Activity or Remission Based on CDAI at Month 12: Tofacitinib vs. IL-6, IPTW
Description: CDAI was a simplified index for assessing disease activity comprising of the SJC, tender/painful joint counts TJC, PtGA and PGA. CDAI is the numerical sum of 4 outcome parameters: SJC and TJC (based on 28-joint assessment range from 0 to 28, higher scores meant worse condition), PtGA and PGA (score range from 0 to 10, assessed on 0-10 cm visual analog scale; higher scores indicated greater affection due to disease activity). CDAI total score = 0 (no disease) to 76 (severe disease), higher scores indicated worse condition. Achievement of LDA was defined by CDAI less than or equal to 10 in participants with moderate or high disease activity CDAI greater than 10 at baseline. IPTW method was used for analysis of this outcome measure.
Time Frame: During 12 month of follow-up post-initiation of tofacitinib or IL-6; retrospective data retrieved, were assembled in this study from 15-May-2024 to 19-July-2024 (approximately 2 months)
Population: as for outcome 1
Measure: Number; unit: Events per 1000 person years
Arm/Group | Tofacitinib | IL-6
Number analyzed (Participants) | 3681 | 2464
Events per 1000 person years | 177.7 | 181.7
Statistical Analysis 1: Comparison: Tofacitinib vs IL-6; Test type: Other; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.79 to 1.09]

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events and all-cause mortality were not planned to be assessed, which explains "at risk" as "0"
Description: Due to non-interventional nature of study, the minimum criteria for reporting an adverse event (i.e., identifiable participant, identifiable reporter, a suspect product, and event) could not be met. Hence, adverse events were not planned to be assessed.
Arm/Group | Tofacitinib | TNFi | Abatacept | IL-6
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-07): https://cdn.clinicaltrials.gov/large-docs/29/NCT06418529/Prot_SAP_000.pdf